CLINICAL TRIAL: NCT03527303
Title: The Impact of 8 Weeks of a Digital Meditation Application on Stress and Job Strain in a Heterogeneous University Employee Cohort
Brief Title: The Impact of 8 Weeks of a Digital Meditation Application on Work Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The University of California's Healthy Campus Network (Other); Headspace, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-23717
Record Dates: First submitted 2018-04-25; First posted 2018-05-17 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Stress, Psychological; Behavioral Symptoms
Keywords: stress; health; meditation; mindfulness; employees; job strain; burnout; work; mood; affect; work related stress
MeSH Terms: conditions — Stress, Psychological; Behavioral Symptoms; Occupational Stress; Burnout, Psychological | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Randomization to either digital meditation condition or wait-list control.
Who Masked: Investigator
Masking Description: Investigator will be blind to condition throughout data accrual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Participants in the intervention group will assigned to a digitally-based meditation intervention (Headspace app- Basics + Stress packs) and asked to use this for at least 10 minutes a day over the course of 8 weeks
  Interventions: Behavioral: Meditation
- Waitlist Control Group (No Intervention): Waitlist control group participants will continue their normal activities and not add any form of meditation during the study period.

INTERVENTIONS:
Behavioral: Meditation — 10 minute per day, 8 week digital meditation
  Arms: Meditation Group

SUMMARY:
The aim of this study is to test the effects of a digital meditation intervention in a sample UCSF employees who report mild to moderate stress. We will randomize UCSF employees to either 8-weeks of a digital meditation intervention (using the commercially available application Headspace) or a waitlist control condition.

DETAILED DESCRIPTION:
The aim of this study is to test the effects of a digital meditation intervention in a sample UCSF employees who report moderate to high stress. We will randomize UCSF employees to either 8-weeks of a digital meditation intervention (using the commercially available application Headspace) or a waitlist control condition.

Participants assigned to the intervention group will be asked to download and use the Headspace mobile application for at least 10 minutes per day for 8 weeks. All study participants will be asked to fill out short (no longer than 25 minutes) questionnaires at baseline, week 4, week 8 (post intervention), and a 4-month follow up period. Among participants who are randomized to the digital meditation intervention, they will also take part in a 1-year follow up. All activities will take place online (via computer or smartphone).

Prior to randomization, participants will go through an eligibility screening and complete the baseline questionnaire battery. The entirety of the study is digital and there are no in-person assessments. Adherence will be tracked remotely. The goal is to recruit as many as 2000 participants (1000 per condition).

ELIGIBILITY:
Inclusion Criteria:

You may join if you:

* Have access to a smartphone or computer every day
* Are fluent in English
* Are a UCSF employee
* Report mild to moderate levels of stress
* Consent: demonstrate understanding of the study and willingness to participate as evidenced by voluntary informed consent and has received a signed and dated copy of the informed consent
* Are at least 18 years of age

Exclusion Criteria:

• You may not join if you are an experienced meditator or have participated in a formal meditation practice in the last 3 months (defined as 3 times per week or more for 10 minutes or more at each practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1458 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress score, as determined by the total score on the Perceived Stress Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Perceived Stress Scale has a total score scale range of 0 to 40, with higher values indicating more perceived stress

SECONDARY OUTCOMES:
Change in job strain, as determined by Siegrist Job Strain Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The job strain measure is a comprised of two sub scales, effort (5 items) and reward (11 items), each ranging from 1 to 4. The job strain score is calculated as the ratio of demand to reward, with a higher ratio reflecting more job strain.
Change in job overcommitment, as as determined by Siegrist Job Strain Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The job overcommitment subscale of the Siegrist Job Strain Scale is comprised of 4 items providing a total score range from 4 to16. A higher total score reflects more job overcommitment.
Change in burnout, as determined by the Bergen Burnout Inventory | Baseline to post-intervention, an anticipated average of 8 weeks
  The Bergen Burnout Inventory is comprised of 9 items, ranging from 1 to 6. The total score range is from 9 to 54 with a higher score reflecting higher burnout.
Change in subjective mindfulness, as determined by total score on Mindful Attention Awareness Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Mindful Attention Awareness Scale is a 15-item measure with each item ranging from a score of 1 to 6. To score the scale, we compute the average score across items, with a higher score reflecting higher levels of mindfulness.
Change in work engagement, as determined by the Utrecht Work Engagement Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Utrecht Work Engagement scale is comprised of 9 items, with a total score ranging from 0 to 54, with higher scores indicating more work engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Aric A Prather, PhD, Principal Investigator — University of California, San Francisco; Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified aggregated data

REFERENCES:
- [Derived] Radin RM, Vacarro J, Fromer E, Ahmadi SE, Guan JY, Fisher SM, Pressman SD, Hunter JF, Sweeny K, Tomiyama AJ, Hofschneider LT, Zawadzki MJ, Gavrilova L, Epel ES, Prather AA. Digital Meditation to Target Employee Stress: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2454435. doi: 10.1001/jamanetworkopen.2024.54435. PMID 39808431